CLINICAL TRIAL: NCT05928858
Title: Clinical And Radiographic Evaluation Of Premixed Bio-ceramic Mineral Trioxide Aggregate Versus Calcium Hydroxide In Indirect Pulp Capping Of Young Permanent Molars: A Randomized Controlled Trial
Brief Title: Clinical And Radiographic Evaluation Of Premixed Bio-ceramic MTA In Indirect Pulp Capping Of Young Permanent Molars
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Adel Abd El-Hafez Osman Hamza, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14422022585603
Record Dates: First submitted 2023-06-24; First posted 2023-07-03 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Indirect Pulp Capping
Keywords: neoputty; premixed bioceramic MTA; young permanent teeth; calcium hydroxide
MeSH Terms: interventions — Calcium Hydroxide; Dycal

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Premixed Bio-ceramic MTA (Experimental): Partial caries removal will be carried out then Premixed Bio-ceramic MTA will be applied as indirect pulp capping agent followed by Glass ionomer filling and composite restoration
  Interventions: Drug: Premixed Bio-ceramic MTA
- Calcium hydroxide (Active Comparator): Partial caries removal will be carried out then calcium hydroxide will be applied as indirect pulp capping agent followed by Glass ionomer filling and composite restoration
  Interventions: Drug: Calcium hydroxide

INTERVENTIONS:
Drug: Premixed Bio-ceramic MTA — Partial caries removal will be carried out then Premixed Bio-ceramic MTA will be applied as indirect pulp capping agent followed by Glass ionomer filling and composite restoration
  Other Names: Neoputty
  Arms: Premixed Bio-ceramic MTA
Drug: Calcium hydroxide — Partial caries removal will be carried out then calcium hydroxide will be applied as indirect pulp capping agent followed by Glass ionomer filling and composite restoration
  Other Names: Dycal, Hydcal
  Arms: Calcium hydroxide

SUMMARY:
The present study aims to evaluate the clinical and radiographic success of premixed bio-ceramic MTA versus calcium hydroxide in indirect pulp capping of young permanent molars.

DETAILED DESCRIPTION:
Researchers are still in search of an ideal material for pulp capping, and they evaluated numerous dental materials. For many decades, calcium hydroxide has been the 'gold standard' material for maintaining pulp vitality. Both clinically and histologically, it has been found to produce satisfactory results in indirect and direct pulp capping because it can stimulate the formation of tertiary dentine by the pulp and it has antimicrobial properties.

Due to the drawbacks of calcium hydroxide, several materials have been developed, such as NeoPUTTY which is premixed bio-ceramic Mineral Trioxide Aggregate (MTA) that triggers hydroxyapatite. Its firm, non-tacky consistency, wash-out resistance, and bioactivity make it a pediatric dentists' preferred material for every pulp need. It also delivers ready-to-use material for immediate placement with zero waste, saving cost and chair time.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have young permanent molars with deep carious lesions.
* Restorable young permanent molars with no clinical symptoms of irreversible pulpitis.
* Permanent molars with no clinical or radiographic signs of pulp necrosis including swelling, fistula, pain on percussion,pathologic tooth mobility, thickening of the periodontal ligament space, radiolucency at the periapical area.

Exclusion Criteria:

* Medically compromised patients who have systemic disease.
* Uncooperative patients who refuse treatment
* Permanent molars that were previously restored
* Children whose parents or caregivers refuse to participate in the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Immediate Postoperative pain | one week
  post operative pain by Verbal analogue scale.It is a 10 cm long horizontal line with points labeled from 0 to 10 where (0) indicates no pain, (1-3) mild pain, (4-6) moderate pain, and (7-10) severe pain.

SECONDARY OUTCOMES:
The thickness of newly formed dentin | 3,6,9,12 month
  The thickness of newly formed dentin will be assessed in Mm through Digora software
Soft tissue pathology | 3,6,9,12 month
  Swelling, sinus tract, fistula, mobility and pain on percussion will be assessed by clinical examination either present or not (binary)
Radiographic changes | 3,6,9,12 month
  Radiolucency at the periapical or furcation area and Internal or external root resorption will be assessed through a digital periapical intraoral radiograph either present or not ( Binary)

CONTACTS AND LOCATIONS:
Overall Officials: Aya Ad Hamza, Phd, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: No
IPD can be shared with citation to the investigator but not personal data of the patients to protect confidentiality.